CLINICAL TRIAL: NCT02963766
Title: A Randomized, Double-Blind Study With an Open-Label Extension Comparing the Effect of Once-Weekly Dulaglutide With Placebo in Pediatric Patients With Type 2 Diabetes Mellitus (AWARD-PEDS: Assessment of Weekly AdministRation of LY2189265 in Diabetes-PEDiatric Study)
Brief Title: A Study of Dulaglutide (LY2189265) in Children and Adolescents With Type 2 Diabetes
Acronym: AWARD-PEDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14171; H9X-MC-GBGC (Other: Eli Lilly and Company); 2016-000361-22 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06-01

CONDITIONS: Type 2 Diabetes
Keywords: Pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo/0.75 milligram (mg) Dulaglutide (Experimental): Participants received placebo administered subcutaneously (SC) for 26 weeks during the double-blind period and open-label 0.75 mg/week dulaglutide for 26 weeks during the Open Label Extension (OLE).
  Interventions: Drug: Dulaglutide; Drug: Placebo
- 0.75 mg Dulaglutide (Experimental): Participants received 0.75 mg/week dulaglutide administered SC for 26 weeks during the double-blind period and open-label 0.75 mg/week for 26 weeks during the OLE.
  Interventions: Drug: Dulaglutide
- 1.5 mg Dulaglutide (Experimental): Participants received 1.5 mg/week dulaglutide administered SC for 26 weeks during the double-blind period and open-label 1.5 mg/week for 26 weeks during the OLE.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
Drug: Placebo — Administered SC
  Arms: Placebo/0.75 milligram (mg) Dulaglutide

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics and pharmacodynamics of the study drug dulaglutide compared to placebo in pediatric participants with type 2 diabetes. The study duration is approximately 60 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes, treated with diet and exercise, with or without metformin and/or basal insulin. Metformin and/or basal insulin dose must be stable for at least 8 weeks prior to study screening.
* Have HbA1c >6.5% to ≤11% at screening visit. If newly diagnosed and not on medicine for diabetes, HbA1c must be between >6.5 % to ≤9%.
* Have a BMI (body mass index) >85 percentile for age, gender and body weight ≥50 kilograms (110 pounds).

Exclusion Criteria:

* Known type 1 diabetes, or positive GAD65 or IA2 antibodies, or history of diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome.
* A history of, or at risk for pancreatitis.
* Self or family history of Multiple Endocrine Neoplasia (MEN) type 2A or B, thyroid C-cell hyperplasia or medullary thyroid cancer, or a blood calcitonin result ≥20 picograms per milliliter (pg/ml) at screening.
* A systolic blood pressure of ≥160 millimeters of mercury (mmHg) or diastolic ≥100 mmHg.
* Active or treated cancer.
* A blood disorder where an accurate HbA1c may not be obtainable.
* A female of childbearing age, sexually active and not on birth control.
* Pregnant or plan to be pregnant during the study, or breastfeeding.
* Taking any diabetic medication other than metformin or basal insulin and have not stopped it 3 months prior to the screening visit (6 weeks for bolus or mealtime insulin).
* Have taken oral steroids within the last 60 days or more than 20 days use within the past year or 1000 micrograms fluticasone propionate per day.
* Using prescription weight loss medications in the last 30 days, or plan to use.
* Taking psychiatric medications for depression or illness or attention deficit hyperactivity disorder (ADHD) if, the doses has changed within the last 3 months.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (23):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Advanced Research Center, Anaheim, California
  - Division of Endocrinology, Diabetes, and Metabolism, Los Angeles, California
  - Childrens Hospital of Orange County, Orange, California
  - Center of Excellence in Diabetes & Endocrinology, Sacramento, California
  - Rady Childrens Hospital - San Diego, San Diego, California
  - JC Cabaccan, San Jose, California
  - Touro University, Vallejo, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Florida Center for Endocrinology & Metabolism, Orlando, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - ECU Pediatric Specialty Care, Greenville, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
  - CAMC Institute, Charleston, West Virginia
- Brazil (8):
  - Instituto Estadual de Diabetes e Endocrinologia, Rio de Janeiro, Rio de Janeiro
  - Centro de Pesquisas em Diabetes, Porto Alegre, Rio Grande do Sul
  - Instituto da Criança com Diabetes, Porto Alegre, Rio Grande do Sul
  - Hospital PUC-CAMPINAS, Campinas, São Paulo
  - Hospital das Clinicas da FMRP, Ribeirão Preto, São Paulo
  - CPCLIN, São Paulo, São Paulo
  - Hospital da Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - UNIFESP - Escola Paulista de Medicina, São Paulo
- France (2):
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hopital Robert Debre, Paris
- Germany (3):
  - Praxis Dr. med. Landers, Mayen, Rhineland-Palatinate
  - Zentrum für klinische Studien, Sankt Ingbert, Saarland
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
- Heim Pal Gyermekkorhaz, Budapest, Hungary
- India (9):
  - Dr Jivraj Mehta Smarak Health Foundation Bakeri Medical Research Centre, Ahmedabad, Gujarat
  - Manipal Hospital, Bangalore, Karmnataka
  - M S Ramaiah Medical College Hospital, Bangalore, Karnataka
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Banaras Hindu University - BHU, Varanasi, Uttar Pradesh
  - Park Clinic, Kolkata, West Bengal
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
- Mexico (6):
  - Health Pharma Professional Research, S.A. de C.V., Mexico City, Federal District
  - Centro de Inv. Medica de Occidente, SC, Zapopan, Jalisco
  - Centro Medico San Francisco, Monterrey, Nuevo León
  - Cli-nica Hospital Cemain, Tampico, Tamaulipas
  - Hospital Angeles Puebla, Puebla City
  - Arke Estudios Clinicos S.A. de C.V., Veracruz
- Centro de Diabetes y Endocrinologia Pediatrica de PR, Bayamón, PR, Puerto Rico
- Saudi Arabia (2):
  - King Saud University Hospital, Riyadh
  - King Salman bin Abdulaziz Hospital - Diabetic Center, Riyadh
- Turkey (Türkiye) (4):
  - Ankara University Medicine Hospital, Ankara, Mamak
  - Sami Ulus Education & Research Hospital, Ankara
  - Duzce University Medical Faculty, Düzce
  - Ondokuz Mayis University Medical Faculty, Samsun
- United Kingdom (2):
  - Alder Hey Children's Hospital, Liverpool, Lancashire
  - St James's University Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.vivli.org/

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Arslanian SA, Hannon T, Zeitler P, Chao LC, Boucher-Berry C, Barrientos-Perez M, Bismuth E, Dib S, Cho JI, Cox D; AWARD-PEDS Investigators. Once-Weekly Dulaglutide for the Treatment of Youths with Type 2 Diabetes. N Engl J Med. 2022 Aug 4;387(5):433-443. doi: 10.1056/NEJMoa2204601. Epub 2022 Jun 4. PMID 35658022
- See also: A Study of Dulaglutide (LY2189265) in Children and Adolescents With Type 2 Diabetes (AWARD-PEDS) — https://trials.lillytrialguide.com/en-US/trial/5RwyJT8t9uI0ISG4U4SEu0

RESULTS

PARTICIPANT FLOW:
Period: Double-Blind Period
Arm/Group | Placebo/0.75 Milligram (mg) Dulaglutide | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Started | 51 | 51 | 52
Received at Least 1 Dose of Study Drug | 51 | 51 | 52
Completed | 47 | 49 | 50
Not Completed | 4 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Withdrawal by Parent or Guardian | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Open Label Extension (OLE)
Arm/Group | Placebo/0.75 Milligram (mg) Dulaglutide | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Started | 47 | 49 | 50
Completed | 45 | 46 | 48
Not Completed | 2 | 3 | 2
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo/0.75 mg Dulaglutide: Participants received placebo administered SC for 26 weeks during the double-blind period and open-label 0.75 mg/week dulaglutide for 26 weeks during the OLE.
- Total: Total of all reporting groups
Arm/Group | Placebo/0.75 mg Dulaglutide | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Total
Number analyzed (Participants) | 51 | 51 | 52 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.20 (2.08) | 14.70 (2.21) | 14.70 (1.81) | 14.50 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 34 | 110
  Male | 10 | 16 | 18 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 31 | 28 | 85
  Not Hispanic or Latino | 25 | 18 | 22 | 65
  Unknown or Not Reported | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 4 | 16
  Asian | 11 | 4 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 5 | 9 | 9 | 23
  White | 25 | 29 | 30 | 84
  More than one race | 3 | 1 | 3 | 7
  Unknown or Not Reported | 0 | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 4 | 7 | 5 | 16
  France | 0 | 2 | 2 | 4
  Germany | 2 | 1 | 0 | 3
  India | 3 | 4 | 4 | 11
  Mexico | 14 | 12 | 10 | 36
  Puerto Rico | 0 | 1 | 1 | 2
  Saudi Arabia | 2 | 0 | 1 | 3
  Turkey | 1 | 1 | 1 | 3
  United Kingdom | 3 | 2 | 0 | 5
  United States | 22 | 21 | 28 | 71
Percentage of Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.14 (1.12) | 7.92 (1.27) | 8.16 (1.39) | 8.08 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (Pooled Doses) at Week 26
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least square (LS) mean in HbA1c was calculated using a restricted maximum likelihood (REML) based mixed-effects model for repeated measures (MMRM) and adjusted by, baseline + insulin Use + metformin Use + treatment + time + treatment*time (Type III sum of squares). Variance-covariance structure = unstructured (for actual value) / unstructured (for change from baseline).
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline HbA1c.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1C
Groups:
- Placebo: Participants received placebo administered SC for 26 weeks.
- Pooled Dulaglutide: Participants received pooled: 0.75 mg/week dulaglutide and 1.5 mg/week dulaglutide administered SC for 26 weeks.
Arm/Group | Placebo | Pooled Dulaglutide
Number analyzed (Participants) | 45 | 100
percentage of HbA1C | 0.5 (0.24) | -0.7 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Pooled Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -1.3, 95% CI 2-sided [-1.8 to -0.7]

2. Secondary Outcome: Change From Baseline in HbA1c (Individual Doses) at Week 26
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS mean in HbA1c was calculated using a REML based MMRM and adjusted by, baseline + insulin use + metformin use + treatment + time + treatment*time (Type III sum of squares). Variance-covariance structure = unstructured (for actual value) / unstructured (for change from baseline).
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- 0.75 mg Dulaglutide: Participants received 0.75 mg/week dulaglutide administered SC for 26 weeks.
- 1.5 mg Dulaglutide: Participants received 1.5 mg/week dulaglutide administered SC for 26 weeks.
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 45 | 50 | 50
percentage of HbA1c | 0.5 (0.24) | -0.5 (0.22) | -1.0 (0.22)
Statistical Analysis 1: Comparison: Placebo vs 0.75 mg Dulaglutide; Test type: Superiority; p = 0.002, Mixed Models Analysis; LS Mean difference (Final Values) = -1.0, 95% CI 2-sided [-1.7 to -0.4]
Statistical Analysis 2: Comparison: Placebo vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -1.5, 95% CI 2-sided [-2.2 to -0.9]

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at Week 26
Description: Fasting blood glucose is a test to determine how much glucose (sugar) is in a blood sample after an overnight fast. Least squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) analysis and adjusted by baseline, strata, treatment, time, treatment*time, (Type III sum of squares). Variance-Covariance structure = Unstructured (for actual value) / Unstructured (for change from baseline). Strata refer to: insulin use + metformin use + baseline HbA1c group [ less than (<) 8%, greater than or equal to (>=) 8%).
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had evaluable fasting blood glucose data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 43 | 49 | 50 | 99
millimoles per liter (mmol/L) | 0.96 (0.45) | -0.47 (0.41) | -1.54 (0.41) | -1.03 (0.29)
Statistical Analysis 1: Comparison: Placebo vs 0.75 mg Dulaglutide; Test type: Superiority; p = 0.021, Mixed Models Analysis; LS Mean difference (Final Values) = -1.44, 95% CI 2-sided [-2.65 to -0.22]
Statistical Analysis 2: Comparison: Placebo vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -2.51, 95% CI 2-sided [-3.72 to -1.29]
Statistical Analysis 3: Comparison: Placebo vs Pooled Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -1.97, 95% CI 2-sided [-3.03 to -0.91]

4. Secondary Outcome: Percentage of Participants With HbA1c ≤7.0%
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: Week 26
Population: All randomized participants who received at least 1 dose of study drug and had evaluable baseline and post-baseline HbA1c.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 45 | 50 | 50 | 100
percentage of participants | 18.42 | 60.00 | 53.19 | 56.52
Statistical Analysis 1: Comparison: Placebo vs 0.75 mg Dulaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.038, 95% CI 2-sided [3.491 to 34.902]
Statistical Analysis 2: Comparison: Placebo vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.666, 95% CI 2-sided [3.653 to 37.253]
Statistical Analysis 3: Comparison: Placebo vs Pooled Dulaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.348, 95% CI 2-sided [4.163 to 30.932]

5. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 26
Description: BMI is an estimate of body fat based on body weight divided by height squared. LS mean were calculated using a MMRM analysis and adjusted by baseline, strata, treatment, time, treatment*time, (Type III sum of squares). Variance-Covariance structure = Unstructured (for actual value) / Unstructured (for change from baseline). Strata refer to: insulin use + metformin use + baseline HbA1c group (< 8%, >= 8%).
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had evaluable BMI data.
Measure: Least Squares Mean (Standard Error); unit: kilograms/square meter (kg/m^2)
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 50 | 51 | 52 | 103
kilograms/square meter (kg/m^2) | -0.0 (0.21) | -0.2 (0.20) | -0.1 (0.19) | -0.1 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 0.75 mg Dulaglutide; Test type: Superiority; p = 0.689, Mixed Models Analysis; LS Mean difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs 1.5 mg Dulaglutide; Test type: Superiority; p = 0.924, Mixed Models Analysis; LS Mean difference (Final Values) = -0.0, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 3: Comparison: Placebo vs Pooled Dulaglutide; Test type: Superiority; p = 0.776, Mixed Models Analysis; LS Mean difference (Final Values) = -0.1, 95% CI 2-sided [-0.6 to 0.4]

6. Secondary Outcome: Percentage of Participants With Self-Reported Events of Hypoglycemia
Description: Summary and analysis of Incidence of all hypoglycemia with Plasma Glucose <54mg/dL.
Time Frame: Week 26
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 51 | 52
percentage of participants | 1.96 | 3.92 | 3.85

7. Secondary Outcome: Percentage of Participants Requiring Rescue for Severe, Persistent Hyperglycemia
Description: Percentage of Participants Requiring Rescue for Severe, Persistent Hyperglycemia was summarized.
Time Frame: Week 26
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 51 | 51 | 52 | 103
percentage of participants | 17.6 | 3.9 | 1.9 | 2.9

8. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Week 26
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 51 | 51 | 52 | 103
participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Pancreatic Enzymes at Week 26
Description: Serum Amylase (total and pancreas-derived) and lipase concentrations were measured.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had evaluable pancreatic enzymes data.
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 47 | 51 | 52 | 103
Units/Liter (U/L)
  Serum Amylase | 0.09 (17.36) | 4.80 (9.39) | 6.50 (8.91) | 5.64 (9.15)
  Serum Amylase, Pancreatic | 0.60 (9.94) | 1.77 (4.72) | 2.90 (6.10) | 2.32 (5.45)
  Serum Lipase | 2.23 (31.99) | 4.37 (8.28) | 3.88 (6.63) | 4.12 (7.47)

10. Secondary Outcome: Number of Participants With Thyroid Treatment-Emergent Adverse Events
Description: Number of Participants with Thyroid Treatment-Emergent Adverse Events were summarized.
Time Frame: Week 26
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 51 | 51 | 52 | 103
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Serum Calcitonin at Week 26
Description: Change from Baseline in Serum Calcitonin was evaluated.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had evaluable serum calcitonin data.
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 47 | 48 | 48 | 96
nanograms per liter (ng/L) | 0.38 (1.70) | 0.28 (0.72) | 0.10 (0.50) | 0.19 (0.62)

12. Secondary Outcome: Percentage of Participants With Allergic, Hypersensitivity Reactions
Description: The percentage of Participants with Allergic and hypersensitivity reactions that were considered possibly related to study drug by the investigator are presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 51 | 51 | 52 | 103
percentage of participants | 2.0 | 3.9 | 1.9 | 2.9

13. Secondary Outcome: Percentage of Participants With Injection Site Reactions
Description: The percentage of participants with at least one treatment-emergent injection site reaction is presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide | Pooled Dulaglutide
Number analyzed (Participants) | 51 | 51 | 52 | 103
percentage of participants | 9.8 | 9.8 | 7.7 | 8.7

14. Secondary Outcome: Number of Participants With Anti-Dulaglutide Antibodies
Description: Dulaglutide anti-drug antibodies (ADA) were assessed at baseline, Weeks 26 and 56. A participant was considered to have treatment-emergent (TE) dulaglutide ADAs if the participant had at least 1 titer that was TE relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline through Week 56
Population: All randomized participants who received at least 1 dose of study drug and had at least one post-baseline Dulaglutide ADA test result.
Measure: Number; unit: participants
Groups:
- Placebo/0.75 mg Dulaglutide: Participants received placebo administered SC for 26 weeks during the double-blind period and open-label 0.75 mg/week dulaglutide for 26 weeks during the open OLE.
Arm/Group | Placebo/0.75 mg Dulaglutide | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 46 | 51 | 52
participants | 3 | 3 | 3

15. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration of Dulaglutide at Steady-state (Cmax,ss)
Description: PK: Maximum Concentration of Dulaglutide at steady-state (Cmax,ss) was derived by a population pharmacokinetics approach. As part of addendum, additional PK samples were taken at week 9.
Time Frame: Week 9: pre-dose,1 to 12 hours post dose and 24 to 96 hours post dose; Week 13: predose and 1 to 12 hours post dose; Week 26: predose; Week 39: up to 2 days postdose; Week 52 and Week 56: PK sample can be taken at any time during the visit
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- 0.75 mg Dulaglutide: Participants received 0.75 mg/week dulaglutide administered SC for 56 weeks.
- 1.5 mg Dulaglutide: Participants received 1.5 mg/week dulaglutide administered SC for 56 weeks.
Arm/Group | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52
nanograms per milliliter (ng/mL) | 31 [28.4 to 33.5] | 62 [56.9 to 67.2]

16. Secondary Outcome: PK: Area Under the Concentration Time Curve Over a 1-week Interval of Dulaglutide at Steady-State [AUC(0-168)ss]
Description: PK: Area Under the Concentration Time Curve over a 1-week interval of Dulaglutide at Steady-State [AUC(0-168)ss] was derived by a population pharmacokinetics approach. As part of addendum, additional PK samples were taken at week 9.
Time Frame: as for outcome 15
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (95% Confidence Interval); unit: nanogram*hour per milliliter (ng*h/ mL)
Arm/Group | 0.75 mg Dulaglutide | 1.5 mg Dulaglutide
Number analyzed (Participants) | 51 | 52
nanogram*hour per milliliter (ng*h/ mL) | 4170 [3770 to 4510] | 8350 [7640 to 9070]

ADVERSE EVENTS:
Time Frame: Up To 56 Weeks
Description: All randomized participants who received at least one dose of study drug. The gender specific events only occurring in male or female participants were adjusted accordingly.
Groups:
- Placebo: Double-Blind Period: Participants received placebo administered SC for 26 weeks.
- 0.75 mg Dulaglutide: Double-Blind Period: Participants received 0.75 mg/week dulaglutide administered SC for 26 weeks.
- 1.5 mg Dulaglutide: Double-Blind Period: Participants received 1.5 mg/week dulaglutide administered SC for 26 weeks.
- Placebo/0.75 mg Dulaglutide: Open Label Extension (OLE): Participants who had received placebo during the double-blind period were given 0.75 mg/week dulaglutide administered SC for additional 26 weeks after the double-blind period.
- 0.75 mg Dulaglutide: OLE: Participants received 0.75 mg/week dulaglutide administered SC for additional 26 weeks after the double-blind period.
- 1.5 mg Dulaglutide: OLE: Participants received 1.5 mg/week dulaglutide administered SC for additional 26 weeks after the double-blind period.
Arm/Group | Placebo: Double-Blind Period | 0.75 mg Dulaglutide: Double-Blind Period | 1.5 mg Dulaglutide: Double-Blind Period | Placebo/0.75 mg Dulaglutide: Open Label Extension (OLE) | 0.75 mg Dulaglutide: OLE | 1.5 mg Dulaglutide: OLE
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/52 | 0/47 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/51 | 1/51 | 1/52 | 0/47 | 1/49 | 2/50
Other Adverse Events (participants affected / at risk) | 26/51 | 25/51 | 28/52 | 18/47 | 16/49 | 20/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: Double-Blind Period (N=51) | 0.75 mg Dulaglutide: Double-Blind Period (N=51) | 1.5 mg Dulaglutide: Double-Blind Period (N=52) | Placebo/0.75 mg Dulaglutide: Open Label Extension (OLE) (N=47) | 0.75 mg Dulaglutide: OLE (N=49) | 1.5 mg Dulaglutide: OLE (N=50)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo: Double-Blind Period (N=51) | 0.75 mg Dulaglutide: Double-Blind Period (N=51) | 1.5 mg Dulaglutide: Double-Blind Period (N=52) | Placebo/0.75 mg Dulaglutide: Open Label Extension (OLE) (N=47) | 0.75 mg Dulaglutide: OLE (N=49) | 1.5 mg Dulaglutide: OLE (N=50)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (4) | 0 (0) | 3 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (8) | 3 (3) | 5 (6) | 2 (2) | 0 (0) | 5 (21)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 8 (13) | 11 (19) | 0 (0) | 1 (1) | 6 (21)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (16) | 8 (13) | 1 (2) | 3 (10) | 6 (12)
Vomiting (Gastrointestinal disorders) | 2 (2) | 9 (10) | 7 (14) | 4 (6) | 4 (4) | 5 (8)
Pyrexia (General disorders) | 2 (2) | 2 (3) | 2 (2) | 2 (3) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (4) | 5 (6) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 2 (3) | 6 (7) | 3 (4) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (8) | 7 (7) | 8 (21) | 2 (2) | 5 (6) | 5 (6)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/41 (1) | 1/35 (1) | 2/34 (4) | 0/38 (0) | 0/34 (0) | 3/34 (3)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/41 (0) | 0/35 (0) | 2/34 (2) | 0/38 (0) | 0/34 (0) | 0/34 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT02963766/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02963766/SAP_001.pdf